CLINICAL TRIAL: NCT05483478
Title: Effectiveness of Combined Mobile Health and Multicomponent Program Intervention on Frailty, Muscle Strength and Health Literacy of the Elderly in the Community
Brief Title: Effectiveness of Mobile Health on Frailty, Muscle Strength and Health Literacy of the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landseed Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hua Chien, Principal Investigator, Landseed Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-018-A2
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Telemedicine; Elderly; Health Literacy
Keywords: mobile health; frailty; health literacy; muscle strength
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile health combined Multi-course Program (Experimental): The experimental group received the combination of mobile health and multi-course intervention. In the pre-test, the experimental group joined the LINE group by scanning the QR code. The LINE messages were nutrition and exercise content, as well as exercise videos. One message each for nutrition and exercise was sent every Monday, Wednesday, and Friday, for a total of 12 weeks. The multi-course includes exercise and nutrition, 1 time per week, 2 hours each time, a total of 12 times, and each unit is 50 minutes long. The three measurement time points of the tracking effect were: before intervention, after 4-times interventions, and after 12-times interventions. The following data were collected in the two groups: frailty assessment, grip strength, lower limb muscle strength, health literacy scale and nutrition knowledge scale.
  Interventions: Combination Product: mobile health combined Multi-course Program
- Multi-course Program (Active Comparator): The control group received multi-course includes exercise and nutrition, 1 time per week, 2 hours each time, a total of 12 times, and each unit is 50 minutes long. The three measurement time points of the tracking effect were: before intervention, after 4-times interventions, and after 12-times interventions. The following data were collected in the two groups: frailty assessment, grip strength, lower limb muscle strength, health literacy scale and nutrition knowledge scale.
  Interventions: Combination Product: mobile health combined Multi-course Program

INTERVENTIONS:
Combination Product: mobile health combined Multi-course Program — mobile health combined Multi-course Program

SUMMARY:
This study explores the effect of mobile health combined with multi-course intervention on frailty, muscle strength, health literacy and nutrition knowledge among the elderly in the community. A longitudinal, repeated test quasi-experimental design was adopted to convenient sampling. Four community care bases in northern Taiwan were selected, and 2 experimental groups and 2 control groups were assigned by computer lottery to participate in the study. 60 in the experimental group and 60 in the control group. The experimental group received the combination of mobile health and multi-course intervention, and the control group only received the intervention of multi-course. The three measurement time points of the tracking effect of the two groups were: before intervention, after 4-times interventions, and after 12-times interventions. The following data were collected in the two groups: frailty assessment, grip strength, lower limb muscle strength, health literacy scale and nutrition knowledge scale. Statistical data were analyzed by SPSS26.0 software. Descriptive statistics include: percentage, mean, standard deviation; inferential statistics include: independent sample t test, chi-square test, generalized estimation model.

DETAILED DESCRIPTION:
The current preventive and delayed disability care programs have problems such as uneven quality, number of participants, and lack of funds. During the COVID-19 epidemic, isolation measures have affected the preventive care of the elderly. More appropriate and innovative service programs should be adopted to expand Promote the prevention and delay of disability care services for the elderly in the community, so that the elderly can actively participate in their own health promotion work, reduce the occurrence of disability, shorten the number of years of disability, and enjoy a high-quality elderly life.

This study explores the effect of mobile health combined with multi-course intervention on frailty, muscle strength, health literacy and nutrition knowledge among the elderly in the community. A longitudinal, repeated test quasi-experimental design was adopted to convenient sampling. Four community care bases in northern Taiwan were selected, and 2 experimental groups and 2 control groups were assigned by computer lottery to participate in the study. 60 in the experimental group and 60 in the control group. The experimental group received the combination of mobile health and multi-course intervention, and the control group only received the intervention of multi-course. The three measurement time points of the tracking effect of the two groups were: before intervention, after 4-times interventions, and after 12-times interventions. The following data were collected in the two groups: frailty assessment, grip strength, lower limb muscle strength, health literacy scale and nutrition knowledge scale. Statistical data were analyzed by SPSS26.0 software includes: percentage, mean, standard deviation; independent sample t test, chi-square test, generalized estimation model.

ELIGIBILITY:
Inclusion Criteria:

* Ability to act independently.
* Conscious and articulate.
* Those who can communicate in Mandarin or Taiwanese.
* Smartphones and Internet access available.
* "LINE" mobile communication software can be used.

Exclusion Criteria:

* Cognitive Impaired Persons.
* mentally illness.
* Those with musculoskeletal injuries of the upper and lower limbs.
* Patients with a history of serious heart and lung diseases.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
frailty assessment | baseline, during the procedure, through study completion
  Study of Osteoporotic Fractures scale was adopted。Include: (1) Weight loss: Loss of 3kg or more in the past without intentional weight loss.
  (2) Weakened lower extremity function: unable to stand up from a chair five times without support by hands.
  (3) Decreased energy: In the past week, did you feel that you couldn't get enough energy to do things? If more than two of the three items are met, frailty is defined; if one is met, the pre-frailty is defined; if not met, no frailty.
muscle strength | baseline, during the procedure, through study completion
  Grip machine。A practice session is given before the test to ensure that the subject understands the test process. The hand grip strength of the elderly in Taiwan is 26 kg for men and 16 kg for women.
Health Literacy | baseline, during the procedure, through study completion
  Mandarin Multidimensional Health Literacy Questionnaire。Each subscale has 4 questions, a total of 20 questions, and each question is scored 1-4 points. After the formula conversion, the score is between 0-50 points. Health awareness level 0-25 is insufficient; 26-33 is limited; 34-42 is sufficient; 43-50 is good.
Nutrition knowledge | baseline, during the procedure, through study completion
  Nutrition knowledge questionnaire。There are 5 true-false questions, 5 multiple-choice questions, a total of ten questions; 1 point for a correct answer, 0 point for a wrong answer, and the score is between 0 and 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Qing-Ping Wu, Doctor, Study Chair — Landseed International Hospital
Locations (1):
- Landseed Intrenational Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No